CLINICAL TRIAL: NCT02583971
Title: Assessment of Thrombotic Status in Patients With Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: East and North Hertfordshire NHS Trust (Other Government)
Collaborators: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Prof Diana Gorog, Professor of cardiology, East and North Hertfordshire NHS Trust
Other Study IDs: No. 1.2 Oct 2015
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Atrial Fibrillation
Keywords: Direct current cardioversion; Medical management; Atrial fibrillation ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole blood Plasma store
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with AF: Split into 3:
  Those patients on treatment for AF involving blood thinning medicines (anticoagulants) +/- heart rate limiting drugs such as B blockers or digoxin. 100 patients in this group.
  Patients undergoing direct current cardioversion (DCCV) to temporarily restore normal (sinus) rhythm. 100 patients in this group.
  Patients undergoing an AF ablation to permanently restore sinus rhythm. 300 patients in this group.

SUMMARY:
Investigators will assess the impact of treatments for atrial fibrillation on participant's thrombotic status

DETAILED DESCRIPTION:
AF affects 1 in 4 people in their lifetime. Although generally thought of as a safe heart rhythm disturbance, the risk associated with AF is through the formation of clot (thrombus) within the heart which be ejected from the heart when it contracts causing a heart attack or perhaps more devastatingly a stroke.

The mainstay of treatment for AF involves thinning the blood with drugs such as warfarin or newer drugs termed novel oral anticoagulants. In addition to this there are 3 main ways of treating the underlying rhythm disturbance:

1. Accept the irregular heart rhythm and simply control the heart rate with heart rate limiting drugs such as beta blockers or digoxin in addition to the blood thinning medicines.
2. Restore the normal heart rhythm with with an electrical shock termed a direct current cardioversion (DCCV). This is usually a temporary measure, indeed 70% of whom will have reverted to AF by 12 months.
3. Attempt to permanently restore sinus rhythm through an atrial fibrillation ablation procedure.

The investigators study, through use of a relatively novel bedside test will examine the effects of each of these management strategies on the thrombotic status of the participant's blood.

Investigators will take blood from in total 500 participants divided between each of the above management strategies which has been decided by their parent teams (i.e. study does not affect their treatment).

Investigators will draw blood from the participants on up to 5 separate occasions over a 12 month period. In the group undergoing a DCCV, blood will be drawn shortly before and after the intervention and at 3 and 12 months post intervention. In the group undergoing an AF ablation blood will be drawn on 5 occasions - the day before the procedure, 1-2 days post, 3-4 days post, 3-4 months post and 12 months post. In the group treated with standard medical therapy, blood will be drawn at the time of enrolment in the study and at 3 and 12 months post enrolment.

It is the investigators hypothesis that permanent restoration of sinus rhythm through an atrial fibrillation ablation procedure will positively affect an individual participant's thrombotic status. There has been recent publication of registry data from the United States suggesting the long term rate of stroke in the population following an AF ablation approaches that of the population who have never suffered AF.

The investigators believe that the cause of the improvement in stroke rates following ablation is an improvement in thrombotic status which we hope to be test for the first time in a powered, prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients aged 18 years or over
2. Patients diagnosed with atrial fibrillation managed in one of the 3 ways outlined above
3. The patient is willing and able to understand the Patient Information Sheet and provide informed consent
4. The patient must agree to comply with the drawing of blood samples for the assessments

Exclusion Criteria:

1. Male and female patients aged < 18 years of age
2. The patient has, in the opinion of the investigator, significant neurological, hepatic, renal, endocrine, gastrointestinal, pulmonary, haemorrhagic, metabolic or other disease likely to confound the study requirements or analyses
3. The patient has a history of substance abuse or demonstrates signs or clinical features of active substance abuse or psychiatric disease
4. Alcohol consumption above recommended safe levels (i.e. more than 21 units per week for males, or more than 14 units per week for females) due to the potential effects of high alcohol levels on platelet reactivity
5. Any illness deemed significant by the investigator during the four (4) weeks preceding the screening period of the study
6. Any major bleeding diathesis or blood dyscrasia (platelets < 70 x 109/l, Hb < 8 g/dl, INR > 1.4, APTT > x 2 UNL, leucocyte count < 3.5 x 109/l, neutrophil count < 1 x 109/l)
7. Currently enrolled in an investigational device or drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population of interest are adults (>18) diagnosed with atrial fibrillation (AF) who will be treated in one of 3 ways:
  1. Medical management
  2. Direct current cardioversion
  3. AF ablation
  In total we aim to sample 500 patients divided into:
  100 - Medical management 100 - Direct current cardioversion 300 - AF ablation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Thrombotic status | 12 months
  This will be assessed using the investigator's novel bedside blood test. Each participant will have blood taken at predetermined points in time over a 12 month period. Some will have blood sampled on 3 different occasions, some on 4 occasions and the majority will have blood sampled on 5 occasions over the 12 months. The Global Thrombosis test provides information of the time taken for whole blood to clot (occlusion time) and then for the clot to naturally break down (lysis time)

SECONDARY OUTCOMES:
Major adverse clinical event (MACE) | 12 months
  Over the time period that investigators are sampling, investigators will also note any major adverse clinical events such as heart attack, stroke or death.

CONTACTS AND LOCATIONS:
Overall Officials: Diana Gorog, MD PhD FRCP, Principal Investigator — East and North Herts NHS Trust